CLINICAL TRIAL: NCT00621556
Title: RG1068 (Synthetic Human Secretin) Enhanced MRCP for Morphological Evaluation of the Known or Suspected Intraductal Papillary Mucinous Neoplasms of the Pancreas
Brief Title: Secretin Enhanced MRCP for Evaluation of the Known or Suspected Intraductal Papillary Mucinous Neoplasms of the Pancreas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor patient enrollment due to logistical issues
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Dr. Dushyant Sahani, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006P002500
Record Dates: First submitted 2008-01-22; First posted 2008-02-22 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Intraductal Papillary Mucinous Neoplasms
MeSH Terms: interventions — Secretin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Drug + MR with MRCP
  Interventions: Drug: RG1068 (Synthetic Human Secretin)

INTERVENTIONS:
Drug: RG1068 (Synthetic Human Secretin) — Dose: 0.2 μg/kg of synthetic human or 18.5 µg for patients over 50 kg Route: Intravenous Frequency: Once Duration: Over 1 minute

SUMMARY:
1. To assess the effect of RG1068 at a dose of 0.2 mcg/kg intravenously (IV) on the diameter of the pancreatic duct when used during Magnetic Resonance Pancreatography
2. To demonstrate that RG1068-enhanced MRCP improves detection and characterization of intraductal papillary mucinous neoplasms (IPMN) relative to unenhanced MRCP in patients with suspected IPMN
3. To correlate findings on MRCP with histologically confirmed malignancy

DETAILED DESCRIPTION:
Until relatively recently, endoscopic retrograde cholangiopancreatography (ERCP) was the primary diagnostic and therapeutic modality for assessing patients with suspected pancreatic disease or abnormalities. However, this invasive procedure carries with it a significant potential for complications including acute pancreatitis, hemorrhage and infection, as well as reactions to contrast material or premedications and exposure to radiation. In addition, the success of such procedures, both from the standpoint of safety and efficacy, is highly dependent on the skill of the endoscopist, and the cost of ERCP is relatively high.

The advent of magnetic resonance imaging has resulted in the development of a less expensive, non-invasive, radiation-free means of assessing the pancreaticobiliary system: Magnetic Resonance Cholangiopancreatography (MRCP). MRCP uses stationary water in biliary and pancreatic secretions as an intrinsic contrast medium, thus facilitating examination of pancreatic and biliary ducts and surrounding tissue. Secretin, which promotes the secretion of pancreatic fluid into the pancreatic ducts, can thereby enhance the MR imaging signal, improving delineation of both normal and abnormal structures, as well as highlighting abnormal fluid collections and leakage. Conversely, filling defects can indicate the presence of stones or mass lesions.

This study is being undertaken to prospectively assess the effectiveness of RG1068-enhanced MRCP relative to unenhanced MRCP for the evaluation of patients with known or suspected IPMN. RG1068 is a synthetic human secretin with a pharmacological profile very similar to that of biological and synthetic porcine secretins. Secretin is a 27-amino acid gastrointestinal peptide hormone that is produced by S-cells in the duodenum in response to the pH decrease caused by the passage of partially digested food from the stomach into the intestine. RG1068 is identical in amino acid sequence to naturally occurring human secretin and differs from porcine secretin in 2 amino acids.

ELIGIBILITY:
Inclusion Criteria:

* Males and females older than 18 years of age
* Is clinically indicated for MRCP of the pancreas based on prior imaging features suggestive or suspicious of IPMN (eg. Cystic lesion in the pancreas along the duct, ductal dilatation)
* Scheduled for MRCP and therapeutic or diagnostic ERCP or surgery for the IPMN
* Has been fully informed and has personally signed and dated the Written Informed Consent and Health Insurance Portability Accountability Act (HIPAA) provisions
* Is a male, or is a female not of childbearing potential, or is a female of childbearing potential who is using effective contraception and has a negative serum pregnancy test on the same day, but prior to, study drug administration
* Is able and willing to complete all study procedures specified in the protocol

Exclusion Criteria:

* Presence of a pancreatic stent
* History of any clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease which, in the opinion of the investigator, precludes study participation
* History of sensitivity to any of the ingredients in the study drug
* Pregnancy
* Any contraindication to MRI procedure, including but not limited to implanted metal devices (e.g., pacemaker, aneurysm clips, cochlear implants)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-02; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
MR & MRCP - Images will be evaluated for quality, main and branch duct visualization, ductal diameter and improved visualization of structural abnormalities with and without use of RG1068. | 1

SECONDARY OUTCOMES:
Laboratory | 2

CONTACTS AND LOCATIONS:
Overall Officials: Dushyant V Sahani, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States